CLINICAL TRIAL: NCT06080412
Title: A Pilot Single-Arm, Multicenter, Prospective, Post-Market 6 Months Follow-Up Clinical Investigation to Evaluate the Safety and Effectiveness of the Blueprint Mixed Reality HOLOBLUEPRINT™ (HOLOBLUEPRINT™).
Brief Title: Blueprint® Mixed Reality Pilot Study
Acronym: BLUEMR
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: UE-03-2022
Record Dates: First submitted 2022-07-06; First posted 2023-10-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Orthopedic Disorder; Arthritis Shoulder; Arthritis, Degenerative; Cuff Tear Arthropathy; Cuff Rotator Full Thickness Tear
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blueprint Mixed Reality HOLOBLUEPRINT™ in Reversed Shoulder replacement: One single cohort of patients receiving a reversed shoulder arthroplasty with the use of Blueprint Mixed Reality HOLOBLUEPRINT™ as per standard of care.

SUMMARY:
A pilot Single-Arm, Multicenter, Prospective, Post-Market 6 months Follow-Up Clinical Investigation to Evaluate the Safety and Effectiveness of the Blueprint Mixed Reality HOLOBLUEPRINT™ (HOLOBLUEPRINT™).

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to assess performance by collecting post-market performance and safety data. Outcome data collected from this pilot clinical investigation will provide descriptive data on performance and safety for Post-Market Surveillance (PMS) reporting, Clinical investigation Reports (CIR), and Clinical Evaluation Reports (CER).

This France-based pilot clinical investigation will include 4 investigating sites.

The sponsors are seeking to enroll 50 subjects undergoing surgery using HOLOBLUEPRINT™. The inclusion period is expected to take approximately 3 months, at an estimated rate of 13 subjects/month.

In case of implant size difference or necessary changes between the preoperative planning and the actual device implanted, the patient will be excluded (Screen Failure) and no analysis will be performed.

Each time an enrolled patient is operated using HOLOBLUEPRINT™, the site must enroll this patient consecutively, assuming the patient meets inclusion/non-inclusion criteria and provides their signed informed consent to participate (according to local requirements). This process of consecutive enrollment is one means of preventing patient selection bias and should strengthen the value of data collected in the pilot clinical investigation.

Data will be collected preoperatively (baseline), during the surgical intervention, and in the immediate postoperative period (no later than 2 weeks postoperative). Then, a 6-month postoperative visit will complete the patient's participation in the pilot clinical investigation. At any time over the course of the clinical investigation, any adverse events will be recorded; both severity and a possible link to the clinical investigation device will be examined.

The device included in the scope of this pilot clinical investigation is commercially available in Europe: Blueprint Mixed Reality HOLOBLUEPRINT™ used in combination with Blueprint Mixed Reality instruments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of the informed consent.
* Informed and willing to sign an informed consent approved by Ethics Committee
* Willing and able to comply with the requirements of the study protocol
* Considered a candidate for on label shoulder arthroplasty using BluePrint™ 3D planning software and shoulder system:

  * Humeral side: Tornier Perform Humeral Stem
  * Glenoid side: Tornier Perform Reversed Glenoid

Exclusion Criteria:

* Inability to comply with the pilot clinical investigation procedures based on the judgment of the assessor (e.g. unable to accurately respond to the pilot clinical investigation questionnaires, and inability to attend the scheduled assessments);
* The subjects belong to a vulnerable group of subjects, including minors, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion (subjects who may not be acting on their initiative) (referred as "vulnerable subject" in the section 3.44 of the ISO 14155 norm);
* Any medical condition that could impact the pilot clinical investigation outcomes' functional significance, at the investigator's discretion (e.g., neuropathy, allergy);
* Bio RSA (Bone graft (Autograft))
* Subject pregnancy;
* Subjects incompatible with Blueprint®'s intended use and CT Protocol (e.g., metallic device close to the shoulder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with shoulder's condition requiring a shoulder surgery with a reversed implants.
  50 patients are planned to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
PERFORMANCE MEASUREMENT: Glenoid Implant Placement Accuracy | 15 days after surgery
  To describe the performance of HOLOBLUEPRINT™ by measuring the difference between postoperative implant placement compared with preoperative simulated implant placement.
  This will be performed using CT scans and a validated internally developed semi-automated software to compare the postoperative images with the preoperative planning.

SECONDARY OUTCOMES:
DURATION OF THE INTERVENTION | Surgery
  Duration of each planning period and of each subsequent surgical intervention.
FUNCTIONAL EVALUATION AT 6 MONTHS (Range of motion) | 6 months after surgery
  Measure the range of motion (in degrees) of the operated shoulder and compare it to the baseline (preoperative) range of motion. Measures will be performed on anonymized photos of patients by an independent central reviewer.
FUNCTIONAL EVALUATION AT 6 MONTHS (ASES Score) | 6 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is based on a 100-point scale that incorporates both pain and function. Higher scores indicate higher quality of shoulder function.
  This assessment will be conducted at the 6-month postoperative visit and compared with the score obtained before surgery
PAIN EVALUATION AT 6 MONTHS (ASES Score) | 6 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is based on a 100-point scale that incorporates both pain and function. Shoulder pain will be analyzed from the pain visual analog scale included in this assessment.
  This assessment will be conducted at the 6-month postoperative visit and compared with the score obtained before surgery
FUNCTIONAL EVALUATION AT 6 MONTHS (Constant score) | 6 months after surgery
  The Constant Score is based on a 100-point scale. It incorporates subjective pain measurements and questions regarding the function of the shoulder with normal daily activities. Higher scores indicate a higher quality of shoulder function.
  This assessment will be conducted at the 6-month postoperative visit and compared with the score obtained before surgery
FUNCTIONAL EVALUATION AT 6 MONTHS (SANE score) | 6 months after surgery
  The Single Assessment Numeric Value (SANE) score is a single-question outcome measure that asks subjects to rate their shoulder function, on a scale of 0 to 100. Higher scores indicate a higher quality of shoulder function.
  This assessment will be conducted at the 6-month postoperative visit and compared with the score obtained before surgery
SAFETY EVALUATION | Up to 6 months after surgery
  Safety measures will be evaluated throughout the patient's participation in the study.
  Adverse events will be evaluated from inclusion to last follow-up and will be documented during the study and categorized as whether they are serious and whether they are related to the study device or procedure.
  The following adverse events will be collected:
  * Adverse Device Effect (ADE)
  * Adverse Event of Special Interest (AESI)
  * Serious Adverse Event (SAE)
  * Serious Adverse Device Effect (SADE)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (4):
- France (4):
  - APHP Ambroise Paré, Boulogne-Billancourt
  - CHU de Brest, Brest
  - Centre Orthopédique Santy, Lyon
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No